CLINICAL TRIAL: NCT01649635
Title: A Phase IV, Multicenter, National, Non-comparative, Open-label Study of Cabazitaxel, Combined With Prednisone and Prophylaxis of Neutropenia Complications in the Second-line Treatment of Patients With Metastatic Castration-resistant Prostate Cancer and After Failure of Docetaxel-based Chemotherapy. Descriptive Assessment of the Circulating Tumor Cells in This Context.
Brief Title: Study of Cabazitaxel Combined With Prednisone and Prophylaxis of Neutropenia Complications in the Treatment of Patients With Metastatic Castration-resistant Prostate Cancer
Acronym: PROSPECTA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABAZ_L_06003; U1111-1123-9025 (Other: UTN)
Record Dates: First submitted 2012-07-20; First posted 2012-07-25 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel; XRP6258; Prednisone; Ciprofloxacin; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cabazitaxel (Experimental): 25 mg/m2, administered as a 1-hour intravenous infusion, on Day 1 of each cycle, every 21 days Prednisone: 10 mg daily throughout the treatment with cabazitaxel Ciprofloxacin: at a dose of 500 mg for 8 days twice daily (total dose 1.0 g) Granulocyte-Colony Stimulating Factors: maximum dose of 600ug for 7 days or until Absolute Neutrophils Count reaches level ≥ 10.000/mm3
  Interventions: Drug: CABAZITAXEL (XRP6258); Drug: Prednisone; Drug: Ciprofloxacin; Drug: G-CSF (Granulocyte colony-stimulating factor)

INTERVENTIONS:
Drug: CABAZITAXEL (XRP6258) — Pharmaceutical form: solution Route of administration: intravenous
Drug: Prednisone — Pharmaceutical form: tablet Route of administration: oral
Drug: Ciprofloxacin — Pharmaceutical form: tablet Route of administration: oral
Drug: G-CSF (Granulocyte colony-stimulating factor) — Pharmaceutical form: solution Route of administration: subcutaneous

SUMMARY:
Primary Objective:

- To assess effectiveness of prophylactic treatment of hematological complications (grade ≥ 3 neutropenia) resulting from cabazitaxel treatment for 21 days after treatment initiation.

Secondary Objectives:

* PSA response rate;
* Descriptive assessment of CTC (circulating Tumor Cells);
* Rates of grade ≥ 3 neutropenia and febrile neutropenia and grade ≥3 diarrhea over the treatment period;
* Description of the Health Quality of Life of the patients;
* Incidence of adverse events.

DETAILED DESCRIPTION:
Screening: 15 days Treatment: until disease progression Post-treatment Follow-up: 12 months

ELIGIBILITY:
Inclusion criteria :

* Histologically proven Castration-Resistant Prostate Cancer (stage IV only);
* Prior failure of treatment with docetaxel; o Documentation of metastasis by imaging.
* Performance status 0 or 1;

Exclusion criteria:

* Previous treatment with chemotherapy, except for docetaxel;
* Previous use of abiraterone;
* Inability to maintain treatment with androgen deprivation if no previous history of orchiectomy;
* Presence of any other active malignancy or history of any tumor diagnosed in the last 5 years, except basal cell or squamous cell carcinoma of the skin or in situ carcinoma of the skin, bladder or anal canal (these tumors do not prevent participation if they have been treated, even in the last 5 years);
* Hypersensitivity or known allergy to any of the treatments under study, including history of severe hypersensitivity reaction (≥grade 3) to docetaxel and/or to polysorbate 80 containing drugs
* History of congestive heart failure or myocardial infarction within the last 6 months, or uncontrolled cardiac arrhythmias, angina pectoris or uncontrolled hypertension;
* Uncontrolled severe illness or medical condition (including uncontrolled diabetes mellitus)
* Presence of severe comorbidity, which in the opinion of the investigator, puts the patient at risk or impairs compliance to the protocol;
* Known seropositivity for HIV;
* Presence of significant psychiatric or neurological disease, in the investigator's opinion;
* Presence of uncontrolled hypercalcemia;
* Refusal to use appropriate contraception during the study period;
* Participation in any clinical trial in the last 12 months, unless there is benefit to the patient to be justified by the principal investigator
* Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5
* Inadequate organ and bone marrow function

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-07; Primary Completion 2014-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with some episode of neutropenia classified as grade ≥ 3 | 21 days

SECONDARY OUTCOMES:
Proportion of patients with episode of neutropenia grade ≥3 | up to 24 months (every 21 days)
Rate of febrile neutropenia | up to 24 months (every 21 days)
Rate of diarrhea grade ≥3 | up to 24 months (every 21 days)
PSA response rate | up to 24 months (every 21 days)
Circulating Tumor Cells Count (CTC) rate | Day 42, Day 84, Day 126 and End of Treatment
Changes from baseline in score derived from the Functional assessment of cancer therapy-prostate (FACT-P) and the Trial Outcome Index (TOI) | up to 24 months (every 21 days)
Number of patients with adverse events | up to 24 months (every 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (6):
- Brazil (6):
  - Investigational Site Number 007, Centro
  - Investigational Site Number 004, Curitiba
  - Investigational Site Number 006, Lajeado
  - Investigational Site Number 005, Porto Alegre
  - Investigational Site Number 001, Santo André
  - Investigational Site Number 002, São Paulo